CLINICAL TRIAL: NCT05517954
Title: Measures of Cortical Excitability in Patients With Post-traumatic Epilepsy, Traumatic Brain Injury Patients Without Epilepsy, and Healthy Controls: a Pilot Study
Brief Title: Cortical Excitability in Post-traumatic Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Collaborators: Alexander Rotenberg, M.D., Ph.D (Unknown)
Responsible Party: Principal Investigator, Pavel Klein, Pavel Klein, MD, Mid-Atlantic Epilepsy and Sleep Center, LLC
Other Study IDs: maesc011
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Brain Injury; Cortical Excitability; Epilepsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects with TBI and PTE: 10 subjects with a history of TBI, diagnosed with PTE (post-traumatic epilepsy). PTE is defined as acquired epilepsy with seizures that developed within ten years of TBI with no other clear cause
- Subjects with TBI, no PTE: 10 subjects with a history of TBI, and absent epilepsy, but TBI in the past two years and any of the following:
  * Multifocal intracerebral hemorrhages (ICH)
  * depressed skull fracture
  * Subdural hematoma (SDH) requiring surgery
  * SDH and ICH
  * Penetrating wound
- Healthy volunteers: 10 healthy volunteers; absent epilepsy or TBI

SUMMARY:
To test whether measures of cortical excitability derived from motor cortex transcranial magnetic stimulation (TMS) in patients with traumatic brain injury reflect heightened excitability relative to healthy controls and whether such measures can be used to distinguish patients with post-traumatic epilepsy from patients with head trauma but no epilepsy

DETAILED DESCRIPTION:
This is a pilot a pilot cross-sectional study to evaluate the utility of TMS-derived biomarkers in PTE prediction and detection. We will measure motor cortex excitability and intracortical inhibition (see below) in TBI patients with PTE (Group 1), TBI patients with average 30% risk of developing PTE who have not yet developed PTE (Group 2) and healthy age- and sex-matched control participants (group 3). 10 adult subjects aged 18-70 will be recruited into each group. We shall obtain a range of TMS metrics in each individual (see below), and, per metric, compare average values among groups by 1-way ANOVA. Our specific hypothesis is that, relative to healthy control, motor cortex TMS measures will indicate increased cortical excitability in participants with PTE, and a trend toward same in patients with TBI who have not developed PTE For subjects in groups 2 and 3, all antiseizure treatments will be stable (unchanged) for 4 weeks prior to evaluation. Subjects will undergo two ppTMS testing separated by 1-2 weeks. Per participant, TMS metrics (see below), will be evaluated for test-retest reliability (our secondary outcome measure)

ELIGIBILITY:
Inclusion Criteria:

Group 1 (N=10):

* Age 18-70
* Sex: male/female
* PTE, defined as acquired epilepsy with seizures that developed within ten years of TBI with no other clear cause
* Stable ASM doses for at least 30 days
* Epilepsy duration for ≥ 6 months

Group 2 (N=10):

* Age 18-70
* Sex: male/female
* Absent epilepsy, but TBI in the past two years and any of the following:

  * Multifocal intracerebral hemorrhages (ICH)
  * depressed skull fracture
  * Subdural hematoma (SDH) requiring surgery
  * SDH and ICH
  * Penetrating wound

Group 3 (N=10):

* Age 18-70
* Sex: male/female
* Absent epilepsy or TBI

Exclusion Criteria:

1. Primary generalized epilepsy
2. Non-epileptic seizures
3. Progressive neurological disease including neoplasm, CNS degenerative disorders including Alzheimer's disease, other forms of dementia
4. Any systemic illness or unstable medical condition that might pose additional risk, including renal or liver disease, clinically uncontrolled cardiac disease, other unstable metabolic or endocrine disturbances, and active systemic cancer
5. Change in dose of any antiseizure medication within 30 days prior to enrollment
6. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators that would interfere with adherence to study requirements;
7. Use of any CNS-active investigational drugs within 1 month of enrollment.
8. Resective epilepsy surgery less than 6 months before study initiation.
9. Implanted electrical device (e.g. vagal nerve stimulator, deep brain stimulator, responsive neurostimulation device, cardiac pacemeaker, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the site's database, plus 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
To compare the cortical excitability in subjects with TBI, TBI with PTE, subjects without TBI and epilepsy | 2-10 years after TBI
  Measures of cortical excitability derived from motor cortex transcranial magnetic stimulation (TMS) in patients with traumatic brain injury reflect heightened excitability relative to healthy controls, and whether such measures can be used to distinguish patients with post-traumatic epilepsy from patients with head trauma but no epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mid-Atlantic Epilepsy and Sleep center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No